CLINICAL TRIAL: NCT03462238
Title: Determinants of Vascular Calcification in Chronic Renal Failure : Impact of Pyrophosphate Levels After Renal Transplantation
Acronym: PyroCal-greffe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-AOI-02
Record Dates: First submitted 2018-01-12; First posted 2018-03-12 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kidney transplant patients (Other): Group of renal transplant patients for 24 months
  Interventions: Procedure: Blood collection for Ppi assay; Radiation: CT Scan
- Dialysis patients (Other): Group of dialysis patients for 24 months
  Interventions: Procedure: Blood collection for Ppi assay; Radiation: CT Scan

INTERVENTIONS:
Procedure: Blood collection for Ppi assay — A 4.5 ml blood sample will be taken with a citrate vacuum tube.
Radiation: CT Scan — A scanner will be performed

SUMMARY:
Arterial calcifications (AC) are constant lesions in patients with Chronic Kidney Diseases (CKD). Renal transplantation would reduce their progression compared to dialysis. AC pathophysiology is a complex and finely regulated process that involves many local and systemic factors, both pro- and anti-calcification. The progression of the CKD is accompanied by an increase in phosphate levels as the renal excretion capacity of inorganic phosphates (Pi) decreases while their digestive absorption remains unchanged. Hyperphosphatremia is a well-identified calcifying factor contributing to ACs in the CKD. On the other hand, pyrophosphate (PPi) is an anti-calcifying factor from the hydrolysis of extracellular ATP by ectonucleotidases. While there are many factors that may contribute to a protective effect against AC progression of renal transplantation, no study has been yet analysed the role of PPi. Plasma concentration of PPi is decreased in dialysis patients compared to non-kidney failure patients.

The main objective of this monocentric, prospective and interventional pilot study will be to compare the progression of CA and [PPi]pl between a group of renal transplant patients over the past 24 months and a group of dialysis patients over the same period of time. The secondary objectives will be to compare the progression of ACs and the ratio[PPi]pl/[Pi]pl between transplanted and dialysis patients. Transplanted patients will be included within 24 (±3) months of transplant. Dialysis patients will be included at 24 (±3) months of the CT scan performed during the pre-transplant check-up. At inclusion, all patients will benefit from a CT scan without injection and a plasma dose of PPi, Pi and other factors involved in controlling calcification.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients for 24 (±3) months or dialysis patients who have performed pre-transplant CT for 24 (±3) months
* Major Patients
* Informed patients who have signed informed consent
* Patients of both sexes
* Patients affiliated to the social security system

Exclusion Criteria:

* Pregnancy in progress (checked by a previous ßHCG pregnancy test)
* Patients whose clinical condition would not allow inclusion in the study.
* Patients not affiliated with social security
* Patients not consenting or unable to understand the protocol and its development
* Progressive cancer pathology
* Patients under guardianship, under curatorship, protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Concentration of plasma PPi | at patient inclusion
Calcification score | at patient inclusion
  The calcification score is based on a computed tomography (CT) scan.

CONTACTS AND LOCATIONS:
Overall Officials: Georges LEFTHERIOTIS, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Pasteur - Unité d'Exploration Fonctionelle Vasculaire, Nice, France